CLINICAL TRIAL: NCT04202224
Title: Pre-emptive Analgesia Effect in Different Psycho-emotional Status Patients During Lower Third Molar Surgical Extractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tomas Puidokas, Practitioner, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5995
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Pre-emptive Analgesia in Different Psycho-emotional Status Patients
MeSH Terms: interventions — Ibuprofen; Acetaminophen; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study (Experimental): Receives pre-emptive analgesia 30min. prior to third molar extraction. NSAID: Ibuprofen 400mg and Acetaminophen 500mg/
  Interventions: Drug: Ibuprofen 400 mg and Acetaminophen 500 mg
- Placebo (Placebo Comparator): Receives glucose tablets as pre-emptive analgesia 30min. prior to third molar extraction.
  Interventions: Drug: Glucose
- Control (Active Comparator): Receives no medication prior to third molar extraction.
  Interventions: Other: No drug

INTERVENTIONS:
Drug: Ibuprofen 400 mg and Acetaminophen 500 mg — Analgesia.
  Arms: Study
Drug: Glucose — Placebo.
  Arms: Placebo
Other: No drug — Standard surgical procedure without any preoperative medication.
  Arms: Control

SUMMARY:
To increase the effectiveness of pain control, it is recommended to use drugs before the pain onset, therefore the pre-emptive analgesia method is considered as a method, which allows decreasing the post-operative pain to minimum. Previous studies evaluated effectiveness of pre-emptive analgesia but no relation to psycho-emotional status was addressed. Our authors believe that the effect of pre-emptive analgesia may vary based on different psycho-emotional status.

45 volunteers who needed extraction of lower third molars were examined and enrolled in the study (study group - 15; placebo - 15; control - 15 volunteers). Ibuprofen 400mg together with 500mg paracetamol was used for pre-emptive analgesia. Difficulty of the operation, heart rate measurements and operation protocol were documented. Surgeon filled his questionnaire after the procedure. Patients on consultation, operation day and 10 days postop. filled a questionnaire which consisted of general, special and pain evaluation sections. Less favorable psycho-emotional status correlated with more severe pain 6h after operation. This relation was mostly expressed in the control group. Psycho-emotional status of placebo patients was accounted for bigger analgesic consumption frequency. Postoperative pain in study group was minimal compared to other groups. Pre-emptive analgesia enhances patient's psycho-emotional status and sustains postoperative pain control during lower third molar surgical extractions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Indications for mandibular third molar removal.

Exclusion Criteria:

* Presence of NSAID usage;
* Acute inflammation in operating site;
* General diseases that might negatively influence the outcomes of operation, such as epilepsy, unstable neurological condition;
* Anticoagulant usage;
* Diabetes mellitus;
* Cardiovascular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Pre-emptive analgesia is effective in a negative psycho-emotional status patients | 4 months
  Pre-emptive analgesia prior to third molard extraction is effective in different psycho-emotional status patients

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian university of health sciences, Kaunas, Lithuania